CLINICAL TRIAL: NCT04675528
Title: A Randomized, Open-label, Two-way Crossover Clinical Trial to Evaluate the Food Effect on Pharmacokinetics and SafEty of DHP107 (Oral Paclitaxel, Liporaxel®) in Patients With Advanced Solid Tumors (FEEL) / EudraCT no : 2020-004976-16
Brief Title: Food Effect on Pharmacokinetics and Safety of DHP107 (Liporaxel®) FEEL Study
Acronym: FEEL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daehwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107CS-7
Record Dates: First submitted 2020-11-23; First posted 2020-12-19 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2022-01

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor; Liporaxel; DHP107; Oral paclitaxel

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, two-way crossover study consisting of two sequences (RT, TR) in patients with advanced solid tumor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting treatment (Experimental)
  Interventions: Drug: DHP107(Oral paclitaxel)
- Fed treatment (Experimental)
  Interventions: Drug: DHP107(Oral paclitaxel)

INTERVENTIONS:
Drug: DHP107(Oral paclitaxel) — DHP107 200 mg/m^2 orally twice daily on Day 1, 8, and 15 in every 28 days (On food effect study day, DHP107 200 mg/m^2 orally once daily on Day 1, 8 of Cycle 1 with fasted or fed condition according to the assigned sequence)
  Other Names: Liporaxel®

SUMMARY:
To evaluate the food effect on pharmacokinetics of DHP107 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are ≥18 years of age on the date of written informed consent.
2. Subjects with histologically or cytologically confirmed advanced solid tumors including but not limited to the listed below for which paclitaxel monotherapy has been determined an appropriate therapy at the investigator's discretion.

   * Angiosarcoma
   * Bladder cancer
   * Breast cancer
   * Cervical cancer
   * Head and neck cancer (if no difficulty with swallowing)
   * Kaposi's sarcoma
   * Lung cancer
   * Ovarian cancer
3. Subjects who have a life expectancy of ≥12 weeks.
4. Subjects who are able to take oral medication.
5. Subjects who have a performance status of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) scale.
6. Subjects who have evaluable disease according to the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST version 1.1).
7. Subjects who have adequate organ functions as indicated by the following laboratory values:
8. Subjects who are willing and able to comply with scheduled visits, treatment plans, laboratory tests, and procedures.
9. Subjects who have voluntarily agreed to participate by giving written informed consent.
10. Women of childbearing potential who have negative pregnancy test results at the screening visit and men with female partners of childbearing potential must agree to use adequate contraception for the duration of the trial and up to 90 days after last dose of study drug

Exclusion Criteria:

1. Subjects who have history of severe hypersensitive reaction to the active ingredient or any excipients of DHP107.
2. Subjects with following surgical history/medical conditions that may affect drug absorption:
3. Subjects who developed cardiovascular disease (unstable angina, myocardial infarction, stroke, and transient ischemic attack) within 24 weeks prior to study entry, which is deemed to be clinically significant by the investigator.
4. Subjects with known active hepatitis B or C infection, or hepatobiliary disease, or known history of immunodeficiency virus infection (However, subjects with Gilbert's Syndrome, asymptomatic gallstones, or stable chronic liver disease are, at the discretion of the investigator, eligible for the study. Subjects who are hepatitis B carriers may be eligible if they are on antiviral therapy 2 weeks prior to study entry).
5. Subjects with neuropathy grade > 2 based on CTCAE v5.0 at the time of study entry.
6. Subjects with uncontrolled medical or mental illness that, in the investigator's judgement, could affect treatment tolerability or compliance.
7. Subjects diagnosed with other malignant primary tumor with an exception of the following:

   * Malignancy diagnosed at least 5 years previously without evidence of recurrence or persistent disease
   * The complete excision of basal/squamous cell carcinoma or papillary thyroid carcinoma or the complete treatment of cervical intraepithelial neoplasia or other in situ carcinoma
8. Subjects with symptomatic or unstable, untreated metastases to the central nervous system (CNS) at the time of screening ('Unstable' means worsening of symptoms within 4 weeks prior to screening).
9. Subjects who are currently receiving alternative cytotoxic agents, regular systemic corticosteroids and medications that could influence drug absorption (e.g. H2-antihistamines, antacids, metoclopramide and charcoal) within 4 weeks prior to entry into the study (C1D1).
10. Subjects who are currently receiving (or unable to stop use the 3 days before the first dose of DHP107 and throughout the study) prescription or non-prescription medications or other products known to be moderate or potent inhibitors/inducers of CYP3A4, P-gp, or CYP2C8.
11. Subjects who cannot intake whole high fat meal offered.
12. Pregnant or breastfeeding women.
13. Subjects who have received any investigational drugs or devices within 4 weeks before the first day of study treatment (C1D1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
• Cmax | Day 1 and Day 8 of Cycle 1(each cycle is 28 days)
  The primary endpoints of this trial are the ratio of geometric means of the following pharmacokinetic parameters following DHP107 administration fed with fasting condition
• Tmax | Day 1 and Day 8 of Cycle 1(each cycle is 28 days)
  and the median difference of the following pharmacokinetic parameters following DHP107 administration fed with fasting condition:

CONTACTS AND LOCATIONS:
Overall Officials: Erika Hitre, M.D., Ph.D, Principal Investigator — National Institute of Oncology
Locations (5):
- Hungary (5):
  - University of Semmelweis, 1st Internal Medicine Clinic, Department of Clinical Pharmacology, Budapest
  - National Institute of Oncology, Budapest
  - University of Debrecen-Clinical Center, Internal Medicine Clinic, Department of Clinical Pharmacology, Debrecen
  - Clinexpert Ltd Phase I. Studycenter, Gyöngyös
  - University of Szeged, Dermatology and Allergology Clinic, Phase I. Investigational site, Szeged